CLINICAL TRIAL: NCT04873336
Title: Tidal Volumes Are Generated Automatically With Closed Loop Ventilation (INTELLIVENT ASV) is Safe in Patients With COVID-19
Brief Title: Closed Loop Ventilation in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Cenk Kirakli, M.D., Professor Doctor Cenk KIRAKLI, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Other Study IDs: IGHCEAH-ICU-5
Record Dates: First submitted 2021-05-04; First posted 2021-05-05 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Covid19; ARDS
Keywords: Mechanical ventilation; Adaptive support ventilation; Transpulnonary pressure; Safety
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intellivent ASV — A closed loop mechanical ventilation mode that adjusts oxygenization and ventilation automatically

SUMMARY:
Transpulmonary pressure may be higher in ARDS patients due to decreased respiratory system compliance. The hypothesis is that tidal volumes which are generated by Intellivent- Adaptive support ventilation (ASV) are safe range by transpulmonary pressure.

DETAILED DESCRIPTION:
Patients will be enrolled in the first 24 hours of admission to the intensive care unit. APACHE-2 and SAPS-2 scores will be noted 24 hours after admission. COVID-19 pneumonia will be confirmed according to World Health Organization (WHO) interim guidance. Level of sedation will be monitored with Ramsey Sedation Scale.

An esophageal balloon will be inserted in order to measure transpulmonary pressure(Ptp). The proper localization will be estimated according to ear-nose-xiphoid length. Localization of the balloon will be confirmed with the Baydur maneuver. Mojoli methods will be used to optimize the balloon filling volume.

All patients will be mechanically ventilated under Intellivent-ASV mode. Initial settings will based on predicted body weight. 45 cmH2O will be determined as target end-tidal carbondiokside (ETCO2) but permissive hypercapnia will be allowed if necessary, to maintain lung protective ventilation. Safe pH value will be determined 7.25 independent from ETCO2 levels in patients who will be applied lung protective ventilation. FiO2 and PEEP will be set to maintain an SpO2 of 88-92%.

Ptpinsp will be calculated by subtracting the esophageal pressure from the alveolar pressure measured during inspiratory pause maneuver. Targeted inspiratory transpulmonary pressure (Ptpinsp) was determined to be below 20 cmH2O. If Ptpinsp exceeds 20 cmH2O, minute-volume (MinVol) will be decreased by 10%. Minvol will be reduced below 100% if necessary, to achieve the target. Expiratory transpulmonary pressure (Ptpexp) will be calculated by subtracting the esophageal pressure from the alveolar pressure measured during expiratory pause maneuver. Targeted Ptpexp was determined from 0 to 3 cmH2O. If Ptpexp is below 0 cmH2O, PEEP will be increased until Ptpexp is positive. If Ptpexp exceed 3 mH2O, PEEP will be decreased until Ptpexp is below 3 mH2O. Transpulmonary pressure will be recorded at the beginning after that at least twice daily morning and evening visits. All measurement will be made in passive condition. Transpulmonary pressure measurement will continue until the patient is awake.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 is confirmed with RT-PCR

  ->18 years of age
* Being intubated less than 24 hours
* Not being planned to be extubated in 24 hours

Exclusion Criteria:

* COVID-19 is not confirmed with RT-PCR
* Having an impaired hemodynamic status
* Esophageal pathologies
* Bronchopleural fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with COVID-19 who received invasive mechanical ventilation due to respiratory failure in intensive care unit
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
Inspiratory Transpulmonary Pressure (Ptpins) | The first 24 hours of mechanical ventilation
  Ptpinsp will be measured with an inspiratory hold maneuver

SECONDARY OUTCOMES:
Expiratory Transpulmonary Pressure (Ptexp) | The first 24 hours of mechanical ventilation
  Ptpexp will be measured with an expiratory hold maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Yildirim, M.D., Principal Investigator — University of Health Sciences, Dr. Suat Seren Chest Diseases and Surgery Training and Research Center
Locations (1):
- 1University of Health Sciences Turkey, Dr Suat Seren Chest Diseases and Chest Surgery Training and Research Hospital, Intensive Care Unit, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No